CLINICAL TRIAL: NCT01500512
Title: GROningen INternational Study on Sentinel Nodes in Vulvar Cancer (GROINSS-V) II: An Observational Study
Brief Title: Observation in Patients With Early-Stage Vulvar Cancer Undergoing Sentinel Lymph Node Dissection
Acronym: GROINSS-V
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Other Study IDs: GOG-0270; NCI-2012-00100 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000721346; GOG-0270; GOG-0270 (Other: NRG Oncology); GOG-0270 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2011-12-24; First posted 2011-12-28 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Stage I Vulvar Cancer; Stage II Vulvar Cancer; Stage III Vulvar Cancer; Vulvar Squamous Cell Carcinoma
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Watchful Waiting

GROUPS / COHORTS (1):
- Observation (observe patients undergoing SLN dissection): Patients receive standard therapy including sentinel lymph node dissection. Patients are then observed to collect information about treatment and outcomes every 2 months for 2 years.
  Interventions: Other: Clinical Observation

INTERVENTIONS:
Other: Clinical Observation — Undergo observation

SUMMARY:
This research trial studies patients with early-stage vulvar cancer undergoing sentinel lymph node dissection. Sentinel lymph node dissection may have fewer side effects than removing all lymph nodes. Observing patients undergoing sentinel lymph node dissection may help doctors confirm the safety of the procedure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To prospectively observe patients who receive radiation +/- chemotherapy immediately after lymph node dissection to confirm the safety of this procedure.

OUTLINE:

Patients receive standard therapy including sentinel lymph node dissection. Patients are then observed to collect information about treatment and outcomes every 2 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have squamous cell carcinoma with a depth invasion > 1 mm
* Patients must have T1 or T2 tumors (International Federation of Gynecology and Obstetrics[FIGO] staging), < 4 cm, not encroaching in urethra, vagina, or anus with clinically negative inguinofemoral lymph nodes
* Localization and size of the tumor are such that peri-lesional injection of the tracers at three or four sites is possible
* Preoperative imaging do not show enlarged (< 1.5 cm) suspicious nodes
* Patients must sign informed consent

Exclusion Criteria:

* Inoperable tumors with diameter > 4 cm
* Patients with inguinofemoral lymph nodes, at palpation clinically suspect for metastases, at radiology enlarged (> 1.5 cm) suspicious groin nodes and with cytologically proven inguinofemoral lymph node metastases
* Patients with multifocal tumors
* Patients who are currently on an investigational drug for the treatment of vulvar cancer are excluded from participation in this trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2012-01-03 (Actual); Primary Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety of sentinel lymph node dissection | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Brian Slomovitz, Principal Investigator — NRG Oncology
Locations (37):
- United States (36):
  - University of Arizona Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Jackson Memorial Hospital-Holtz Children's Hospital, Miami, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Baystate Medical Center, Springfield, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Morristown Medical Center, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
- Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada